CLINICAL TRIAL: NCT02437799
Title: Analysis of Changes in the Pulse Oximeter Waveform and Blood Pressure During Spinal Anaesthesia for Caesarean Section: an Observational Study
Brief Title: Dicrotic Notch and Hypotension at Caesarean Under Spinal Anaesthesia
Acronym: DINOCS
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH18900
Record Dates: First submitted 2015-04-01; First posted 2015-05-08 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Hypotension
Keywords: Pulse oximeter; Caesarean section; hypotension; Spinal anaesthesia
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Caesarean section spinal anaesthesia: Dicrotic Wave analysis of pulse oximeter of Women undergoing planned caesarean section under spinal anaesthesia.
  Interventions: Other: Dicrotic wave analysis

INTERVENTIONS:
Other: Dicrotic wave analysis — We will download data from the pulse oximeter that is being used to monitor the patient during their surgery.

SUMMARY:
BACKGROUND:

Hypotension occurs commonly during spinal anaesthesia for caesarean section and may result in detrimental effects to the mother and foetus. A previous pilot study where images of the pulse oximeter waveform study were taken, found that the dicrotic wave moved away from the systolic wave during the onset of hypotension.

AIMS:

The investigators wish to download electronic data which describe the pulse oximeter pulse wave to more accurately assess movement of the diastolic wave relative to the systolic wave during spinal anaesthesia for caesarean section.

METHODOLOGY:

20 women undergoing caesarean section under spinal anaesthesia will be recruited by informed consent for this observational study. Data downloaded from the pulse oximeter will be analysed to identify movement of the dicrotic wave relative to the systolic wave and this will be related to changes in blood pressure.

EXPECTED OUTCOMES:

The investigators will establish best way to analyse changes in the pulse oximeter waveform and the relationship between changes in pulse oximeter waveform morphology and the onset of hypotension during spinal anaesthesia for caesarean section.

IMPLICATIONS:

Analysis of movement of the dicrotic wave could be used to anticipate and thus avoid severe hypotension during spinal anaesthesia for caesarean section.

DETAILED DESCRIPTION:
BACKGROUND:

When a baby is delivered by a surgical procedure (a caesarean section) the women will usually have a spinal anaesthetic. With a spinal anaesthetic local anaesthetic is injected into the spinal fluid to make the woman numb from her chest to her feet allowing her to be comfortable but awake during the birth. One of the common side effects of a spinal anaesthetic is that the woman's blood pressure may fall making her feel unwell and (rarely) causing stress to the unborn baby.

During a caesarean section the blood pressure is usually measured every few minutes using a cuff around the upper arm. However, the blood pressure may fall too quickly to be detected in a timely fashion by this intermittent means. One of the other monitors used in all cases is called a pulse oximeter. When this is attached to the patient's finger it detects the pulse rate and how much oxygen there is in the blood. The pulse oximeter also produces an image of the pulse wave in the finger. There is one pulse wave for every time the heart beats and it has two components. The main part of the wave (the systolic wave) is caused by the heart beat and the second part of the wave (the dicrotic wave) is a result of some of the energy from the heart beat bouncing back from blood vessels.

In a previous study we used a digital camera to take images of the pulse oximeter monitor screen so that we could record changes in the shape of the pulse wave. We found that as patients' blood pressure fell the dicrotic wave moved further away from the systolic wave. We now intend to down load the electronic data that make up the pulse oximeter waveform, so that we can analyse the changes that occur more accurately.

We believe that falling blood pressure may be detected earlier using analysis of movement of the dicrotic wave than by our standard monitoring. This is because currently blood pressure is measured intermittently whereas the pulse oximeter waveform is displayed continuously. Drugs could then be given promptly to stop the blood pressure from falling so low that the woman feels unwell or the unborn baby is affected.

AIMS:

Our aim is to observe changes in the position of the dicrotic wave during spinal anaesthesia for caesarean section and relate these to the occurrence of low blood pressure.

METHODOLOGY:

Following ethical approval 20 women undergoing caesarean section under spinal anaesthesia will be recruited by written informed consent. In theatre the electronic data which describe the pulse oximeter waveform will be downloaded by means of a data logger. In parallel, we will manually record the other perioperative data including the blood pressure. We will then use the data to establish the best way of accurately and reproducibly identifying the dicrotic wave when it moves in relation to the onset of low blood pressure. As this is an observational study, the management of the case will be at the discretion of the attending anaesthetist in discussion with the patient and will not be altered by inclusion in the study.

EXPECTED OUTCOMES:

1. We will establish the best way to detect movement of the dicrotic wave.
2. We will establish the temporal relationship between movement of the dicrotic wave and fall in blood pressure during spinal anaesthesia for caesarean section.

IMPLICATIONS:

Anaesthetists will be able to use movement of the dicrotic wave to anticipate and avert low blood pressure during spinal anaesthesia for caesarean section.

ELIGIBILITY:
Inclusion Criteria:

Patients with an uncomplicated pregnancy presenting for elective caesarean section under spinal anaesthesia where surgery and anaesthesia are anticipated to be uncomplicated.

Exclusion Criteria:

Conditions which may impair the ability of the technology to read accurately such as:

* Reduced peripheral perfusion e.g. Raynaud's phenomenon
* Circulating pigments e.g. bilirubin
* Nail varnish that cannot be removed Diseases of pregnancy: e.g. pregnancy induced hypertension Significant co-existing maternal disease - e.g. congenital heart disease Inability to speak fluent English

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women undergoing planned caesarean section under spinal anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
1. To download electronic data which describe the pulse oximeter pulse wave to accurately assess movement of the diastolic wave relative to the systolic wave during spinal anaesthesia for caesarean section. | Data will be downloaded for approximately 20 minutes
  Data will be collected during planned caesarean section under spinal anaesthesia

SECONDARY OUTCOMES:
Time course of cardiovascular changes | twenty minutes
  1. To clearly document the time-course of cardiovascular changes and hypotension during spinal for caesarean section
Preliminary cardiovascular data | twenty minutes
  2. To provide preliminary data to characterise cardiovascular changes during hypotension
Vascular behaviour | twenty minutes
  4. To characterise changes in vascular behaviour, and to determine their time course, before and after onset of hypotension and the given treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ian Wrench, MBChB,FRCA, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield NHS Trust, Sheffield, South Yorkshire, United Kingdom